CLINICAL TRIAL: NCT02833883
Title: A Phase 1b Study of Enzalutamide Plus CC-115 in Men With Castration-Resistant Prostate Cancer (CRPC)
Brief Title: Use of an Experimental Drug, CC-115, With Enzalutamide in Men With Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-074; c15-160 (Other: Prostate Cancer Clinical Trials Consortium, LLC (PCCTC))
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer; Castration Resistant Prostate Cancer
Keywords: Enzalutamide; CC-115; 16-074
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; 1-ethyl-7-(2-methyl-6-(1H-1,2,4-triazol-3-yl)pyridin-3-yl)-3,4-dihydropyrazino(2,3-b)pyrazin-2(1H)-one

ARMS (1):
- Enzalutamide plus CC-115 (Experimental): The first several study participants will receive the lowest dose. If the drug does not cause serious side effects, it will be given to other study participants at a higher dose. The doses will continue to increase for every group of study participants until the maximum tolerated dose is identified. Participants at each site will participate in the dose escalation phase of the study. During the dose escalation phase, study participants will be assigned sequentially to three dose levels in groups (cohorts) of 3 to 6 subjects per dose level: Cohort 1: CC-115 at 5 mg dose twice a day & enzalutamide at 160 mg once a day. Cohort 2: CC-115 at 10 mg dose twice a day & enzalutamide at 160 mg once a day. The protocol has been amended to accrue an additional in the expansion phase treated at 7.5 mg BID. Amended to treat expansion group with 5mg BID of CC-115.
  Interventions: Drug: Enzalutamide; Drug: CC-115

INTERVENTIONS:
Drug: Enzalutamide
Drug: CC-115

SUMMARY:
The main purpose of this study to define the good and/or bad effects of the combination of enzalutamide and CC-115 in patients with castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and HIPAA authorization for the release of personal health information.

NOTE: HIPAA authorization may be either included in the informed consent or obtained separately.

* Males 18 years of age and above with a life expectancy of at least 6 months.
* Histological or cytological proof of prostate cancer
* Willing to provide a tumor sample via biopsy from a metastatic site of disease to be collected at screening if safe and feasible per treating investigator discretion. Adequate archival tissue can be used if available in lieu of baseline biopsy.
* Documented progressive metastatic CRPC based on at least one of the following criteria:

  * Rise in PSA: a minimum of 3 rising levels, with an interval of at least 1 week between each determination. The last determination must have a value ≥1 ng/mL, obtained within 4 weeks of starting study drug
  * Measurable disease: new or progressive soft tissue disease on computerized tomography (CT) or magnetic resonance imaging
  * Radionuclide bone scan: at least 2 new bone lesions, as defined by the Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria33
* Serum testosterone < 50 ng/dL. Patients must continue primary androgen deprivation with an LHRH analogue (agonist or antagonist) if they have not undergone orchiectomy
* ECOG performance status of 0-1
* Finasteride, bicalutamide and nilutamide discontinued at least 4 weeks prior to registration.
* Physiologic doses of corticosteroids are permitted (i.e., no more than 10mg of prednisone daily).
* At least 4 weeks must have elapsed from the use of palliative radiation, Strontium-89, Radium-223, or approved immunotherapy prior to registration.
* Less than or equal to 5 half lives or 4 weeks, whichever is shorter, from the use of any investigational therapy prior to registration.
* Normal organ function with acceptable initial laboratory values within 14 days of registration.

  * ANC ≥ 1,500/μl
  * Hemoglobin ≥ 9g/dL
  * Platelet count ≥ 100,000/μl
  * Creatinine ≤ 1.5 x the institutional upper limit of normal (ULN), or 24-hr clearance ≥50 mL/min
  * Potassium ≥ 3.5 mmol/L (within institutional normal range, or correctable with supplements)
  * Bilirubin ≤ 1.5 x ULN (unless documented Gilbert's disease)
  * SGOT (AST) ≤ 2.5 x ULN
  * SGPT (ALT) ≤ 2.5 x ULN
  * Glycated hemoglobin (HbA1c < 6.4%
* Able to take oral medication without crushing, dissolving or chewing tablets.
* Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Prior exposure to enzalutamide, ARN-509, or other investigational AR-directed therapy
* Prior exposure to abiraterone acetate, ketoconazole or other specific CYP-17 inhibitors
* Prior exposure to agents specifically targeting both mTOR complexes (dual TORC1+TORC2 inhibitors) and/or PI3K/AKT pathways
* Prior chemotherapy for castration resistant disease. Chemotherapy given in the castration-sensitive setting is permissible. At least 6 months from registration must have elapsed since chemotherapy was last received.
* Symptomatic central nervous system metastases
* Known history of acute or chronic pancreatitis
* Persistent diarrhea or malabsorption ≥ NCI CTCAE Grade 2, despite medical management
* Clinically significant cardiac diseases, including any of the following:

  * Unstable angina pectoris
  * Myocardial infarction ≤ 3 months prior to registration
  * Other clinically significant heart disease such as congestive heart failure requiring treatment or uncontrolled hypertension
* Uncontrolled diabetes mellitus
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
* Major surgery ≤ 2 weeks prior to registration or who have not recovered from side effects of such therapy. Subjects must have recovered from any effects of recent radiotherapy that might confound the safety evaluation of study drug.
* Hematopoietic stem cell transplant ≤ 3 months prior to registration.
* Adults of reproductive potential not employing two forms of birth control:

  * Males having partners who are female with child-bearing potential must agree that they and/or their partners will use at least two effective contraceptive methods (including one barrier method) when engaging in reproductive sexual activity throughout the study from the time of informed consent, and will avoid conceiving for 28 days after the last dose of CC-115.
* Known human immunodeficiency virus (HIV) infection
* Known chronic hepatitis B or C virus (HBV/HCV) infection
* Concurrent active second malignancy for which the subject is receiving therapy, other than non-melanomatous skin cancer or superficial transitional cell carcinoma.
* History of seizure or any condition that may predispose to seizure including, but not limited to, underlying brain injury, stroke in the past 6 months, primary brain tumors, brain metastases
* Active treatment with medications that lower the seizure threshold which cannot be held:

  * Aminophylline/theophylline;
  * Atypical antipsychotics (e.g., clozapine, olanzapine, risperidone, ziprasidone);
  * Bupropion;
  * Lithium;
  * Pethidine;
  * Phenothiazine antipsychotics (e.g., chlorpromazine, mesoridazine, thioridazine);
  * Tricyclic and tetracyclic antidepressants (e.g., amitriptyline, desipramine, doxepin, imipramine, maprotiline, mirtazapine).
* Any other condition which, in the opinion of the Investigator, would preclude participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
establish the maximum tolerated dose (MTD) | 1 year
  Subjects will be treated in cohorts of size three and six and the dosage will be escalated if the clinical toxicity is acceptable. The maximum tolerated dose is defined as the highest dose level with an observed incidence of DLT in no more than one out of six subjects treated at a particular dose level. A DLT will be determined by cycle 1 toxicity, although all-cycle toxicity will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Rathkopf, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - University of California San Francisco, San Francisco, California
  - John Hopkins Medical Center, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Washington School of Medicine, Seattle, Washington

REFERENCES:
- [Derived] Zhao JL, Antonarakis ES, Cheng HH, George DJ, Aggarwal R, Riedel E, Sumiyoshi T, Schonhoft JD, Anderson A, Mao N, Haywood S, Decker B, Curley T, Abida W, Feng FY, Knudsen K, Carver B, Lacouture ME, Wyatt AW, Rathkopf D. Phase 1b study of enzalutamide plus CC-115, a dual mTORC1/2 and DNA-PK inhibitor, in men with metastatic castration-resistant prostate cancer (mCRPC). Br J Cancer. 2024 Jan;130(1):53-62. doi: 10.1038/s41416-023-02487-5. Epub 2023 Nov 18. PMID 37980367
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/